CLINICAL TRIAL: NCT01229579
Title: Effect of Zinc Supplementation on Response to Oral Polio Vaccine in Infants in Pakistan: a Randomized, Controlled Trial
Brief Title: Effect of Zinc Supplementation on Response to Oral Polio Vaccine in Infants in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Founding Director, Centre of Excellence in Women and Child Health, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1291-Peds/ERC-09
Record Dates: First submitted 2010-10-25; First posted 2010-10-28 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Poliomyelitis
Keywords: poliomyelitis; OPV; zinc supplement; diarrhea; placebo; double blind randomized control trial; elemental zinc; seroconversion; bOPV; infants; immunity
MeSH Terms: conditions — Poliomyelitis; Diarrhea; HIV Seropositivity | interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zinc Supplement (Experimental): 2.5 ml Zinc supplement syrup daily containing 10 mg of elemental zinc
  Interventions: Drug: Zinc Sulfate
- Placebo (Placebo Comparator): 2.5 ml supplement syrup daily without elemental zinc
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Zinc Sulfate — 2.5 ml Zinc supplement syrup daily containing 10 mg of elemental zinc from day 14 to 18 weeks of age.
  Arms: Zinc Supplement
Other: Placebo — 2.5 ml placebo syrup daily with containing no elemental zinc from day 14 to 18 weeks of age.
  Arms: Placebo

SUMMARY:
Pakistan is one of the 4 developing countries where cases of poliomyelitis are still being identified. Despite the incessant efforts by WHO and UNICEF, this disease is far from control. There is a need to develop new and innovative strategies to contain the disease and eradicate it from the countries where new cases continue to be identified.

Zinc is an essential component of scores of enzymes in the human body. Recent reports have indicated that this trace element along with other micronutrients enhances the protective functions of immune cells. Moreover, zinc deficiency leads to dysregulation of balanced host responses to infection resulting into decreased antibody production and suppressed immunity. Zinc is also an essential cofactor for thymulin which is known to modulate cytokine release and induce immune cell proliferation. Zinc deficiency is also found to impair an individual's epithelial barrier function, which may further depress the vaccine entry into the mucosal cells.

Role of zinc in the prevention of diarrheal diseases and other infections in children is well documented. However, there are very few reports about its contribution to enhanced immunity by supporting body's natural defense system.

Zinc insufficiency is widespread in socioeconomically deprived children in South Asia and the recent most national nutrition survey (2003) . Moreover, diarrhea is also very common in infants in Pakistan. Such diarrheal episodes can limit entry of attenuated polio virus into the mucosal cells, thereby, leading to inadequate immune response. Association between recent diarrheal history and increased vaccine failure in infants has been shown in a study from Brazil. The recent Lancet Nutrition series has also recommended regular zinc supplementation to address child undernutrition and stunting and underscored the need to treat diarrheal episodes with zinc to expedite recovery. Other recent studies of zinc supplementation in low birth weight infants in South Asia have also shown significant improvement in diarrheal disease burden and mortality.

On the basis of these lines of evidence, it is possible that some of the cases of vaccine failure in this region could be a consequence of compromised immunity and, hence, diminished response to OPV. This could potentially be reversed by addressing such gross undernutrition and micronutrient deficiencies. It can thus be hypothesized that zinc supplementation at community scale would enhance the immune response in infants to OPV.

In order to test this research question, the investigators propose to undertake 12-month randomized controlled trial among a cohort of Pakistani infants of 0-14 days of age. Such a trial would enable us to understand the synergistic role of zinc (if any) with OPV in enhancing immune response against polio and sero-conversion rates.

DETAILED DESCRIPTION:
The investigators propose to carry out a randomized controlled clinical trial in Pakistan to assess the efficacy of zinc supplementation in the first 18 weeks of life on seroconversion due to OPV.

Infants of 0-14 days of age will be recruited and randomized into 2 groups; all the groups would receive the respective OPV doses according to the EPI schedule, and the intervention group, in addition, would receive 10 mg of elemental zinc on a daily basis, for 18 weeks, starting at the age of 14 days.

At 18 weeks (after the 4 weeks of last OPV), the investigators provide an additional dose of bOPV as a challenge and collect stool samples to at 0 and 7 days after delivery at of the bOPV.

Study settings The rural settlement of Hala (population ~ 200,000), located about 200 km north-east of Karachi, Pakistan would be the selected study site, as a high proportion of at-risk under 5 children reside in the area. The large proportion of this population falls in the lower socioeconomic group, according to a recently conducted census in 2008, making the site eminently suitable to test out the trial hypotheses.

The Department of Pediatrics & Child Health, AKU has established liaison with the community members and local government stakeholders, with its research office located in a district-level tertiary care hospital. The nearby vaccination center would assist in delivering the OPV doses, according to the EPI schedule, along with other EPI vaccines. The tertiary health care center (Taluka Hospital, Hala) would provide a place for evaluation and treatment for any unforeseen adverse reactions / events, free of cost.

Study population The trial would recruit full term healthy infants of either sex at or soon after birth and randomize them for supplementation as soon as possible after birth (within 72 hours and in tandem with the first OPV dose). Infants beyond this age and preterm infants (< 37 weeks gestation or < 2 kg birth weight) would be excluded.

Sampling strategy Eligible subjects would be identified and randomized to the respective intervention and comparative groups using computer generated three cell block randomization permutation tables.

Group A: Standard OPV schedule and oral zinc supplement (as 10 mg zinc sulfate liquid preparation) daily for 18 weeks.

Group B: Will receive standard OPV schedule and standard care. An identical placebo preparation, similar in taste, color and consistency will also be administered daily for 18 weeks.

The groups would receive standard OPV doses at birth, at 6 weeks, at 10 weeks and at 14 weeks of age, as recommended by the expanded program of immunization (EPI). As practiced by WHO and UNICEF, OPV doses would also be administered in the cohort, through the polio mass vaccination campaign, scheduled twice in every 3 months. The zinc and placebo preparation will be administered in equal volumes (2.5 ml daily), prepared by Atco Laboratories Limited, one of the leading pharmaceutical industries in Pakistan. . They would hold the allocation codes, replenish supplies at fortnightly intervals and maintain consumption records. The research and monitoring staff will be fully blinded to these preparations.

Given the need to follow individual level response, the investigators have chosen an individual randomized trial as opposed to a cluster randomized trial. The investigators shall employ a computerized block randomization strategy with groups matched in blocks of 20, with the codes maintained by Atco Laboratories Limited and the Chair of the AKU ERC.

Trained field workers will visit the households, 2 times a week to assess compliance to the assigned intervention at their respective time schedules, motivate families and evaluate the child as per a standard format. For the recruits in the research study, incentives would be provided in the form of soaps and cloths to be provided when the field teams visit the household for collection of blood samples from the study subjects. These have been selected in view of the immediate need of these to the recruited child residing in the area of Hala and through years of formative research for comparable projects in rural Sindh. These incentives have deliberately been kept modest so as not to pose undue incentives for participation. The health workers would replenish zinc or placebo supplies every 12 days (in 30 ml bottles).

Enrollment of participants Sample size estimates There is scarcity of research indicating the seroconversion rates to OPV among infants residing in a rural population of Pakistan. The investigators assumed that a conservative estimate of seroconversion to OPV among infants till 14 weeks of age for a rural population of Pakistan would be about 50%. These seroconversion rates are consistent with the lower limits of OPV seroconversion rates observed among breastfed young infants in one solitary study on the subject in Pakistan. To detect a 20% improvement in seroconversion rates upon zinc administration, the investigators would require a minimum of 242 subjects (121 subjects occupying each group) at 5% level of significance and 90% power. Estimating a 30% maximum dropout or refusal rate in comparable studies involving serological testing, the investigators would require a total of 320 subjects, with 160 subjects occupying each group.

Identification and informed consent A cohort of pregnant women (in their third trimester) would be identified through the baseline census and subsequent updates during the surveillance period. The investigators will then identify births within 24 hours of birth through an information system employing the assistance of Lady Health Workers (LHWs) of the area and the traditional birth attendants (TBAs). Families will be visited prior to birth to sensitize them about the study and provide an information sheet. Following notification of births, the families will be visited again and informed consent sought prior to initial randomization. The recruited infants and families will be visited, 3 times per week to assess morbidity and growth (height, weight, mid-arm circumference and head circumference). Close liaison would be maintained with the local vaccination centers, where the OPV doses would be administered to the infants according to the EPI schedule of Immunization. Efforts would be made by the research staff to maintain a record of all vaccinations of the recruited cohort, along with dates for subsequent vaccinations.

Surveillance and data collection A research team would be assembled, constituting of research supervisors, field supervisors, research medical officers, phlebotomists and community health workers.

For the census update, a data collector is capable of visiting at least 30 households per day; thus the census update could be covered in a months' time.

Recruitment of subjects in the trial could get covered in less than 2 months. For the trial activity, at least 8 teams would be delegated, with each covering at least 40 households per day. Each household (bearing one potential subject) would be visited 2 times in a week.

A 3-day training program would be imparted to familiarize them of the research protocol, the field operations for the activities of the census/survey and the research trial and measures for completing the forms. A series of data collection forms would be drafted (initially in English; then translated to Urdu and Sindhi languages) to collect information during the entire research period. A case recruitment form (CRF) would be drafted, which would be filled by research medical officers and would bear questions/items on birth history, immunization status, medical history, anthropometry and physical examination. The subjects would be followed up on a regular basis (2 times a week) by the research appointed community health workers with a minimum qualification of matriculation (grade 10 education), using a pre-defined follow up form. The CHWs will record data on immunization status, medical history and management of any ailment (especially diarrhea), anthropometric assessment and medical examination, and laboratory test results (blood serology and ELISA). Immunization status of each recruit would be maintained for every OPV dose provided to the recruited infants. The data would be collected by the CHWs during their regular follow ups in the area through assessment of vaccination records and finger marking during or after campaigns. A supplementation form would be maintained regularly to ensure compliance in all groups and replenished. This would be recorded by the community health workers undertaking household surveillance. All the forms would bear the general information of the child and the intervention codes allotted by Atco laboratories. Research medical officers, in addition to leading the field teams, would also be entrusted to oversee any untoward events/reactions, among the study subjects. These would be brought to their notice by the circulating CHWs. If encountered, the adverse events would be documented followed by its clinically appropriate treatment. If a child, outside the recruited cohort is identified as in need of health care, the CHWs may refer the child to the Taluka Hospital, Hala.

Laboratory Analysis Blood samples (approximately 3 ml from the cubital fossa of either arm) would be collected at birth, at 6 weeks and at 18 weeks of age of the recruited infant, by phlebotomists with relevant experience of drawing blood among infants. The blood samples would be analyzed for polio seroconversion rates. Neutralizing antibodies would be determined using the methods recommended by WHO [9]. The investigators will evaluate antibody responses to OPV by serotype in close collaboration with CDC (Atlanta). A subset of the samples will also be locally tested by ELISA to determine the sensitivity and specificity of ELISA as compared to the gold standard neutralization assays in detecting polio antibodies.

In order to investigate the impact of zinc on immune response to OPV, the investigators would determine the status of zinc (serum levels) in infants in all the groups. These would be determined from blood samples collected at birth, at 6 weeks and at 18 weeks of age and analyzed using atomic absorption spectrophotometry using established micromethods. Other micronutrient indicators influencing systemic and mucosal immunity (hemoglobin, ferritin and vitamin A) would also be analyzed from the collected blood specimens of the recruited subjects.

The blood samples would be collected from the field and transported to the Nutrition Research Laboratory, Department of Pediatrics & Child Health, AKU. A transport mechanism is well established which brings the blood and other biological samples from Hala/Matiari field site to the main laboratory at AKU on a daily basis. To save costs the same mechanism would also be employed for transportation of blood samples to the Research Laboratory at AKU.

Study duration The study is expected to last in total for 12 months; initial 3 months for census activities and field preparation and training activities, 6 months for the actual research trial, inclusive of recruitment, intervention, follow up and laboratory tests and the last 3 months for finalization of data analyses and preparation of the final report.

In addition, the investigators will collect stool samples to at 0 and 7 days after delivery at of the bOPV. The stool samples would be collected from the field and transported to the National Institute of Health (NIH), Pakistan and processed according to the standard protocol used in the global polio laboratory network, including poliovirus isolation, ITD and sequencing. Non-polio enterovirus (NPEV) will be isolated but not characterized. A transport mechanism is well established which brings the stool and other biological samples from Hala/Matiari field site to the Aga Khan University on a daily basis, where the samples will be stored until shipment to the NIH (a WHO Regional Polio Network Laboratory) in Islamabad.

Study variables

* Outcome variables: Seroconversion rates of polio virus (type 1 and type 3), from blood samples collected at the time of recruitment, at 6 weeks and 18 weeks, and prevalence of excretion of poliovirus serotypes 1, 3 at 0 and 7 days after the administration of bOPV
* Other variables: Data would be collected on birth history, immunization status, medical history and management, number and rates of diarrheal episodes, breast feeding practices, laboratory nutritional indices, anthropometric measurements (weight for age, weight for height and height for age), physical examination and vital signs, and other laboratory parameters, like serum zinc, C-reactive protein, polio virus seroconversion rates, etc.

Statistical analyses The collected data would be dual entered in a data base developed using Foxpro, and for further analysis using Statistical Package for Social Sciences (SPSS) version 18 (SPSS Inc., Chicago, IL).

Frequencies for continuous variables would be expressed as means ± standard deviations. Proportions would be calculated for categorical outcomes. Means would be compared using paired t-test. Chi square tests of independence would be employed for determining differences in associations. Differences in seroconversion rates and prevalence of excretion, if any, would be evaluated using ANOVA and non-parametric tests. Multiple logistic regression analysis will be undertaken to determine the nature of relationship between serum zinc status and optimal vaccine seroconversion.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 14 days of healthy newborns

Exclusion Criteria:

* Infants beyond 14 days of age
* Preterm infants (< 37 weeks gestation or < 2 kg birth weight).

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates of polio virus (type 1 and type 3), from blood samples collected at the time of recruitment, at 6 weeks and 18 weeks. | From birth to 18 weeks

SECONDARY OUTCOMES:
Prevalence of excretion of poliovirus serotypes 1, 3 at 0 and 7 days after the administration of bOPV | 18 and 19 Weeks
Effect of zinc supplementation on growth of infants | Day 14 to 18 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Project Office, Aga Khan University, Matiari, Matiari, Sindh, Pakistan